CLINICAL TRIAL: NCT02106611
Title: Tissue and Functional Assessment of Myocardial Injury in Hodgkin Lymphoma (HL) Survivors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 14-017
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hodgkin Lymphoma Survivor
Keywords: MRI; stress echo; Clinical Assessment; 14-017

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hodgkin Lymphoma Survivor: This is a prospective cross-sectional study of 200 HL survivors whose treatment included mediastinal RT at initial diagnosis or relapse, and are at least 5 years from last HL treatment.
  Interventions: Other: Clinical Assessment; Procedure: Stress cardiac MRI; Procedure: Stress echocardiogram

INTERVENTIONS:
Other: Clinical Assessment — HL treatment will be determined by review of available medical records as archived at MSKCC. Recorded variables will include: (1) RT - field, fractional and cumulative dose, and duration; (2) chemotherapy - regimen, planned interval, dose per cycle, and cumulative dosages. Patients will also be asked to complete the FACT-LYM questionnaire and the FACIT Fatigue questionnaire.
Procedure: Stress cardiac MRI — Both imaging tests will be performed within a 30 day interval, with the two modalities interpreted by dedicated study investigators blinded to the results of the other modality.
Procedure: Stress echocardiogram — Both imaging tests will be performed within a 30 day interval, with the two modalities interpreted by dedicated study investigators blinded to the results of the other modality.

SUMMARY:
This study will test whether cardiac MRI can improve early detection of Hodgkin lymphoma associated heart disease compared to a stress echocardiogram. By doing both stress echocardiography and cardiac MRI, we will compare the ability of the two tests to detect heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Classical or nodular lymphocyte predominant HL treated at Memorial Sloan-Kettering Cancer Center.
* Age ≥ 18 years
* Treatment for HL that included mediastinal RT at initial diagnosis or relapse.
* ≥ 5 years from last HL treatment.

Exclusion Criteria:

* Primary HL diagnosis prior to 1980.
* Additional mediastinal RT or subsequent cardiotoxic systemic therapy for secondary malignant neoplasm.
* Known CAD/CHF (defined as documented myocardial infarction, cardiac revascularization, angiographic obstructive CAD, or decreased LV function [EF < 55%] during prior clinical care).
* Contraindication to MRI (i.e. pacemakers, defibrillators, or aneurysm clips, or other implanted ferromagnetic objects), gadolinium (i.e. known hypersensitivity to gadolinium, advanced renal insufficiency as defined by glomerular filtration rate <30 ml/min/1.73m^2).
* Contraindication to exercise stress testing other than the above (i.e. unstable angina or severe valvular stenosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2026-02-06 (Actual); Study Completion 2026-02-06 (Actual)

PRIMARY OUTCOMES:
compare the prevalence of cardiac injury | 2 years
  detected by cardiac MRI to that detected by stress echocardiography among a broadly representative cohort of Hodgkin lymphoma survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/